CLINICAL TRIAL: NCT03947645
Title: Intensive Neurorehabilitation and Stimulation in Chronic Stroke Patients With Severe Motor Impairment of the Upper Extremity
Brief Title: Intensive Neurorehabilitation and Stimulation in Chronic Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: In-Tens
Record Dates: First submitted 2019-05-02; First posted 2019-05-13 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Chronic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ipsilesional stimulation (Experimental): Ipsilesional stimulation
  Interventions: Device: Ipsilesional stimulation
- Contralesional stimulation (Experimental): Contralesional stimulation
  Interventions: Device: Contralesional stimulation

INTERVENTIONS:
Device: Ipsilesional stimulation — Device: ipsilesional transcranial stimulation, neuromuscular Stimulation over target muscle
  Arms: Ipsilesional stimulation
Device: Contralesional stimulation — Device: contralesional transcranial stimulation, neuromuscular stimulation over target muscle
  Arms: Contralesional stimulation

SUMMARY:
Chronic stroke patients (> 6 months) with severe motor impairment of the upper extremity will be enrolled in this single-centre, randomized controlled clinical trial (RCT). All patients will take part in two blocks of high-intense motor training with concurrent neuromuscular stimulation of the paretic upper extremity. In a randomized, cross-over block design, patients will receive transcranial stimulation of either the ipsi- or contralesional hemisphere.

DETAILED DESCRIPTION:
Chronic stroke patients (> 6 months) with severe motor impairment of the upper extremity and non-proportional recovery will be enrolled in this single-centre, randomized controlled clinical trial (RCT). All patients will take part in two blocks of high-intense motor training with concurrent neuromuscular stimulation of the paretic upper extremity. In a randomized, cross-over block design, patients will receive transcranial stimulation of either the ipsi- or contralesional hemisphere.

The primary outcome measure is the Fugl-Meyer Assessment for upper extremity (FM-UE), acquired at baseline, after the intervention period, and at 3 months follow-up. Secondary outcome measures consist of further clinical parameters and biomarkers of corticospinal connectivity.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Chronic stage of stroke (> 6 months)
* No active finger extension/hand opening of the paretic side

Exclusion Criteria:

* Pregnancy
* Epilepsy
* Metal implants
* Pacemaker

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (Upper Extremity) | change from baseline to both directly after intervention and 3 months after

SECONDARY OUTCOMES:
Action Research Arm Test (ARAT) | change from baseline to both directly after intervention and 3 months after
  Motor Impairment of the upper extremity. Several objects in different sizes and weights should be moved by patients.
Arm-A | change from baseline to both directly after intervention and 3 months after
  Questionnaire on capability to care for the paretic arm in different situations of daily living. Scale ranges from 0 (no problems) to 4 (impossible to do).
Modified Ashworth Scale (MAS) | change from baseline to both directly after intervention and 3 months after
  Spasticity in different body parts. Scale ranges from 0 (no spasticity) to 4 (rigid).
Fugl-Meyer Assessment (Lower Extremity) | change from baseline to both directly after intervention and 3 months after
  Assessment of motor impairment of the lower extremity.
10m walking test | change from baseline to both directly after intervention and 3 months after
  Assessment of motor impairment of the lower extremity.
National Institute of Stroke Scale (NIHSS) | baseline
  Assessment of severity of stroke and neurological deficits. Scale ranges from 0 (normal) to 2, 3 or 4 (depending on the item).
Modified Rankin Scale (mRS) | change from baseline to both directly after intervention and 3 months after
  Degree of disability after stroke on a scale from 0 (no symptoms) to 6 (dead).
EQ-5D | change from baseline to both directly after intervention and 3 months after
  Questionnaire on subjective health status. Patients should rate their health status for that day in different tasks of daily living on a scale from no problems, minor problems, moderate problems, big problems to not possible at all.
CAHAI-13 | change from baseline to both directly after intervention and 3 months after
  Test on activities of daily living. Patients should perform several tasks and are scored from 1 (total assist) to 7 (complete independence).
Stroke Impact Scale | change from baseline to both directly after intervention and 3 months after
  Questionnaire on subjective impact of stroke on daily living and health status. Scale ranges from 1 (most negative answer) to 5 (most positive answer).
Barthel Index | change from baseline to both directly after intervention and 3 months after
  Questionnaire on extent to which patients can perform activities of daily living on their own. Patients can reach 0 (cannot perform any task) to a maximum of 100 points (can do everything on their own).
Hospital Anxiety and Depression Scale | change from baseline to both directly after intervention and 3 months after
  Questionnaire on anxiety and depression. Scale ranges from 0 (most positive answer) to 3 (most negative answer).
Neurological Fatigue Index | change from baseline to both directly after intervention and 3 months after
  Questionnaire on fatigue in the last two weeks. Scale ranges from no agreement at all, no agreement, agreement to some extent to full agreement.
NEO-Fünf-Faktoren Inventar | baseline
  Personality questionnaire with 60 statements that patients should rate ranging from strong disagreement, disagreement, neutral, agreement to strong agreement.
Situational Motivation Scale | change from baseline to both directly after intervention and 3 months after
  Questionnaire on motivation to participate in training. Scale ranges from 0 (not correct at all) to 6 (strongly agree).
Berlin Social Support Scale | change from baseline to both directly after intervention and 3 months after
  Questionnaire to evaluate social support. Patients should rate different questions regarding their most important attachment figure ranging from no agreement at all, no agreement, agreement to some extent to full agreement.
Credibility/Expectancy Questionnaire | change from baseline to both directly after intervention and 3 months after
  Questionnaire to evaluate expectancies on current program. Scale rangs from 0 (most negative) to 9 (most positive).

OTHER OUTCOMES:
Elektroencephalography in resting and active states | change from baseline to both directly after intervention and 3 months after
Input-Output curves and motor maps with transcranial magnetic stimulation | change from baseline to both directly after intervention and 3 months after
Task-related and evoked electromyography | change from baseline to both directly after intervention and 3 months after
Camera and marker-based motion capturing | change from baseline to both directly after intervention and 3 months after

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tübingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided